CLINICAL TRIAL: NCT02205931
Title: A Randomised Controlled Trial of the Ketogenic Diet in the Treatment of Epilepsy in Children Under the Age of Two Years
Brief Title: Ketogenic Diet in Infants With Epilepsy (KIWE)
Acronym: KIWE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Alder Hey Children's NHS Foundation Trust (Other); Bristol Royal Hospital for Children (Other); Birmingham Women's and Children's NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); Sheffield Children's NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Lancashire Care NHS Foundation Trust (Network); Newcastle-upon-Tyne Hospitals NHS Trust (Other); St George's University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/0656
Record Dates: First submitted 2013-12-16; First posted 2014-08-01 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Ketogenic diet; Antiepileptic drugs; Randomised controlled trial
MeSH Terms: conditions — Epilepsy | interventions — Diet, Ketogenic; Carbamazepine; Clobazam; Clonazepam; Ethosuximide; Lamotrigine; Levetiracetam; Nitrazepam; Phenytoin; rufinamide; Valproic Acid; stiripentol; Topiramate; Vigabatrin; Zonisamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketogenic diet (Experimental): 8 week trial of the ketogenic diet (KD) therapy. Children allocated to KD therapy will have their diets individually calculated by a paediatric dietitian with consideration of daily calorie requirements, adequate protein intake for growth and vitamin and mineral supplementation. All diets will be implemented according to a classical KD protocol, i.e. based on a ratio of fat to carbohydrate and protein that will usually be between 2:1 and 4:1.
  Interventions: Other: Ketogenic diet
- Antiepileptic drug therapy (Active Comparator): The control intervention will be drug therapy with the most appropriate further antiepileptic drug (AED) for a particular child, depending on their presenting seizures and syndrome and previous drugs used, and chosen by the expert clinician responsible for management of the patient's epilepsy according to a standardised manual (consensus document) written following the initial workshop of the paediatric neurologists from all the trial centres.
  Interventions: Drug: Antiepileptic drug therapy

INTERVENTIONS:
Other: Ketogenic diet — The ketogenic diet is a high fat diet designed to mimic the effects on the body of starvation. The premise is the main energy intake is fat, which is utilised in the body and produces ketones.
  Arms: Ketogenic diet
Drug: Antiepileptic drug therapy — The control intervention will be drug therapy with the most appropriate further antiepileptic drug for a particular child, depending on their presenting seizures and syndrome and previous drugs used, and chosen by the expert clinician responsible for management of the patient's epilepsy.
  Other Names: Carbamazepine; Clobazam; Clonazepam; Ethosuximide; Lacosmide; Lamotrigine; Levetiracetam; Nitrazepam; Phenytoin; Rufinamide; Sodium Valproate; Stiripentol; Topiramate; Vigabatrin; Zonisamide
  Arms: Antiepileptic drug therapy

SUMMARY:
Epilepsy, a condition where individuals are prone to recurrent epileptic seizures, is the most common chronic neurological disorder in children. Epilepsy onset is most common in the first two years of life and is associated with poor prognosis for seizure control and neurodevelopmental outcome.

The ketogenic diet (KD) is a medically supervised diet that is high in fat and restricted in carbohydrates and protein. KD therapy has shown to be an effective treatment for seizures in children with epilepsy older than two. Associated benefits include: a reduced requirement for routine and emergency antiepileptic drugs (AED) and fewer seizure related hospital admissions. Although reports suggest that KD therapy improves seizures in younger children there is no high quality trial data that demonstrates effectiveness and safety in this age group. The KD is resource intensive, requiring dietetic and physician time; data is required to justify expansion of services to cater for the apparent need.

The investigators therefore propose a prospective multicentre randomised trial to investigate the effectiveness and safety of the KD in children with epilepsy under the age of 2, who have failed to respond to two or more AEDs. Children will be randomly assigned to either receive the KD or further AEDs. The allocated treatment will be started after a 2week baseline period, and it's effectiveness assessed after 8 weeks. Seizure diaries will be used to record seizures and related events, a questionnaire will be used to assess diet tolerance; also growth and blood biochemistry will be monitored.

The information obtained from this study is necessary to optimise choices in epilepsy treatment, aiming to improve outcomes and thus determine whether and when the KD should should be used.

DETAILED DESCRIPTION:
The project proposed is a randomised controlled multicentre study of infants with epilepsy who have failed to respond to two or more pharmacological treatments (antiepileptic drugs (AEDs) or corticosteroids), comparing ketogenic diet to treatment with a further AED.

Children for this study will be recruited from 8 paediatric neurology centres in the South of England who have an established KD service for children with epilepsy. The collaborating paediatric neurologists based in these centres are named co-applicants on this proposal. All children ages 3 to 24 months will be considered if they have a diagnosis of epilepsy, namely continuing seizures despite a trial of 2 or more AEDs (including corticosteroids) and are experiencing at least 8 seizures a week.

Children will be excluded if they are shown to have: a metabolic disease contradicting the use of KD; a progressive neurological disease; severe gastrooesophageal reflux or have undergone a previous failed trial of KD. In addition, families should be able to attend clinic on the required timeline. KD meal plans will be accurately calculated for each child individually by a dietitian with consideration of daily calorie requirements, fat to carbohydrate ratio (3:1 or 4:1), adequate protein intake and vitamin and mineral supplementation. Ongoing adjustments to the diet by the dietitian are determined by weight gain and the degree of ketosis.

1. Baseline assessment: Written consent will be obtained from eligible children. Full history including seizure type, neurological examination, weight, length and head circumference will be documented. Randomisation to KD or standard AED group will be carried out with the support of the UCL PRIMENT Clinical Trials Unit (CTU).

   Investigations to be performed in the KD group (or if clinically indicated in the AED group) will include FBC, U&Es, Glucose, LFTs, Calcium, Magnesium, Phosphate, Zinc, Selenium, Acylcarnitine profile, Cholesterol, Triglycerides, Urate, 25 hydroxy Vitamin D, urine calcium/creatinine, urine organic acids. An EEG will be performed if clinically indicated.
2. Observation period of 2 weeks: No changes of regular AEDs. Emergency seizure treatments will continue as required( acute treatment with benzodiazepines). The following data will be recorded in a standardized diary (these data will continue to be recorded throughout the intervention period of 8 weeks): seizure types, seizure frequency, number of emergency seizure treatments required, contacts with the NHS due to seizure exacerbation (hospital admissions number of days, A&E and or GP attendances)
3. Start of the classical KD or further AED. The classical KD will be administered as per protocol of the treating service. The recording of seizure types and frequency is to be continued.
4. Second Assessment (4 weeks after the start of the treatment period, all patients): clinical review including weight; documentation of seizure frequency, and tolerability of the diet in randomised KD group by questionnaire.
5. Third/final assessment (8 weeks after starting treatment/all patients). Clinical review including neurological examination, weight, length and head circumference. Documentation of seizure outcome (from seizure diaries). KD group only: completion of tolerability questionnaire, blood investigations (FBC, U&Es, Glucose, LFTs, plasma bicarbonate, calcium, magnesium, phosphate, zinc, selenium, acylcarnitine profile, cholesterol, triglycerides, urate, nonesterified fatty acids, blood ketones) and urine calcium/creatinine ratio. EEG will be performed if clinically indicated.

Dependent on seizure response, KD (diet group) or AED (standard AED group) will then be continued or changed. Those in the AED group of failed will be offered KD outside the context of the trial. It would be anticipated that clinical data would be collected on all patients to 12 months to determine retention rates.

Exit criteria: Children will withdraw from the treatment prior to 8 weeks should there be q >50% increase in seizure frequency from the baseline, or if intolerable side effects are not resolved by manipulation of KD or medication. A safety monitoring committee will be convened.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 month and 24 months of age (not beyond second birthday at baseline).
2. Diagnosis of epilepsy confirmed.
3. At least an average of 4 seizures/week in baseline period.
4. Failed response to previous trial of two anti-epileptic drugs. In the case of infantile spasms this could include a trial of corticosteroids.
5. Children with written informed consent from parent/guardian.

Exclusion Criteria:

1. Age <1m or > 24 months of age
2. No secure diagnosis of epilepsy
3. < 4 seizures/week on average in baseline period
4. Trial of < 2 AEDs
5. Continues on corticosteroids in previous 3 months prior to randomisation
6. Metabolic disease contraindicating use of the ketogenic diet e.g. pyruvate carboxylase deficiency, MCAD from previous medical investigation and screening at baseline.
7. Progressive neurological disease
8. Severe gastroesophageal reflux
9. Previous treatment with the ketogenic diet
10. Concurrent participation in another clinical trial of an investigational medicinal product.
11. Patients who are prescribed AEDs not listed in the trial IMPs

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of seizures | 6 - 8 weeks
  Number of seizures experienced during weeks 6 - 8

SECONDARY OUTCOMES:
Responder rate | 8 weeks
  number of children seizure free and relationship between medium chain fatty acids and seizure control

OTHER OUTCOMES:
Retention on treatment | 12 months
  retention on treatment, quality of life and neurodevelopmental outcome

CONTACTS AND LOCATIONS:
Overall Officials: Helen Cross, FRCP(UK), Principal Investigator — UCL Institute of Child Health
Locations (11):
- United Kingdom (11):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Lancashire Teaching Hospitals NHS Foundation Trust, Lancashire
  - Leeds Teaching Hospital, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Sheffield Children's NHS Foundation Trust, Sheffield

REFERENCES:
- [Derived] Titre-Johnson S, Schoeler N, Eltze C, Williams R, Vezyroglou K, McCullagh H, Freemantle N, Heales S, Kneen R, Marston L, Martland T, Nazareth I, Neal E, Lux A, Parker A, Agrawal S, Fallon P, Cross JH. Ketogenic diet in the treatment of epilepsy in children under the age of 2 years: study protocol for a randomised controlled trial. Trials. 2017 Apr 26;18(1):195. doi: 10.1186/s13063-017-1918-3. PMID 28446244